CLINICAL TRIAL: NCT01635803
Title: Comparing the Effectiveness and Costs of Bevacizumab to Ranibizumab in Patients With Retinal Vein Occlusions (The BRVO Study)
Brief Title: Comparing the Effectiveness and Costs of Bevacizumab to Ranibizumab in Patients With Retinal Vein Occlusions (BRVO)
Acronym: BRVO
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Leiden University Medical Center (Other); Free University Medical Center (Other); Erasmus Medical Center (Other); Radboud University Medical Center (Other); UMC Utrecht (Other); University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Prof. dr. R.O. Schlingemann, Clinical Professor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL35869.018.11
Record Dates: First submitted 2012-06-28; First posted 2012-07-10 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Retinal Vein Occlusion
Keywords: bevacizumab; ranibizumab; retinal vein occlusions; randomized clinical trial; Macular edema
MeSH Terms: conditions — Retinal Vein Occlusion; Macular Edema | interventions — Bevacizumab; Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ranibizumab (Active Comparator): Monthly injections with ranibizumab during 6 months
  Interventions: Drug: Ranibizumab
- Bevacizumab (Active Comparator): Monthly injections with bevacizumab during 6 months
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — 1.25 mg bevacizumab administered by monthly interval for six months (6 injections).
  Other Names: Avastin
  Arms: Bevacizumab
Drug: Ranibizumab — 0.5mg ranibizumab administered by monthly interval for six months (6 injections).
  Other Names: Lucentis
  Arms: Ranibizumab

SUMMARY:
The primary objective is to demonstrate the non-inferiority of bevacizumab in the treatment of patients with macular edema secondary to a retinal vein occlusion (branch or central) as determined by the change in best-corrected visual acuity in the study eye from baseline to month 6.

DETAILED DESCRIPTION:
Objective: to compare the effectiveness and costs of 1.25 mg bevacizumab to 0.5 mg ranibizumab, given as monthly intravitreal injections during 6 months.

Study Design: This will be a randomized, controlled, double masked, clinical trial in 296 patients in 7 academic trial centres in The Netherlands.

Study population: patients older than 18 years of age with macular edema secondary to a retinal vein occlusion and a best corrected visual acuity (BCVA) score between 78 and 20 letters in the study eye.

Outcomes: The primary outcome measure will be the change in BCVA in the study eye from baseline to month 6.

Secondary outcomes will be amongst others the proportion of patients with a gain of 15 letters or more and/or a BCVA of 20/40 or more at 6 months and the costs per quality adjusted life-year of the two treatments

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients > 18 years of age with vision loss due to foveal center-involved ME secondary to branch or central retinal vein occlusion diagnosed within 6 months before study initiation, who have signed an informed consent;
* BCVA equal or more than 24 and less or equal to 78 letters in the study eye at screening using ETDRS- like visual acuity testing charts at a testing distance of 4 meters
* Mean central subfield thickness more than 275 micron on 2 OCT measurements.

Exclusion Criteria:

1. Women of child-bearing potential.
2. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive serum pregnancy test (human chorionic gonadotropin > 5 mIU/ml);
3. Inability to comply with study procedures;
4. Active intraocular inflammation in either eye at enrolment;
5. Any active infection in either eye at the time of enrolment;
6. History of uveitis in either eye at any time;
7. Structural damage within 600 micron of the center of the macula in the study eye likely to preclude improvement in visual acuity following in the resolution of macular edema, including atrophy of the retinal pigment epithelium, subretinal fibrosis, laser scar(s), epiretinal membrane involving fovea or organized hard exudate plaques;
8. Uncontrolled (neovascular) glaucoma in the study eye at screening. (IOP > 24 mmHg on medication or according to investigator's judgment);
9. Evidence of vitreomacular traction in the study eye;
10. Patients who are monocular or have a Snellen VA in the non-study eye ≤ 1/300 at visit 1;
11. Any intraocular surgery in the study eye within 3 months prior to randomization;
12. Planned medical or surgical intervention during the 6-months study period;
13. Panretinal laser photocoagulation in the study eye within 3 months prior to or during the study;
14. Focal/grid laser photocoagulation in the study eye 3 months prior to study entry;
15. Treatment with anti-angiogenic drugs in the study eye within 3 months prior to randomization;
16. Use of other investigational drugs at the time of enrolment, or within 3 months or 5 half-lives from enrolment, whichever is longer;
17. History of intravitreal corticosteroids in study eye within 4 months prior to randomization;
18. Ocular conditions in the study eye that require chronic concomitant therapy with topical ocular or systemically administered corticosteroids;
19. History of stroke or transient ischemic attack (TIA) within 6 months prior to enrolment;
20. History of myocardial infarction within 3 months prior to randomization;
21. Current use of or likely need for systemic medications known to be toxic to the lens, retina or optic nerve, including deferoxamine, chloroquine/hydroxychloroquine (Plaquenil), tamoxifen, phenothiazines and ethambutol;
22. Known hypersensitivity to fluorescein, bevacizumab or ranibizumab or any component thereof or drugs of similar chemical classes;
23. Any type of advanced, severe or unstable disease or its treatment, that may interfere with primary and/or secondary variable evaluations including any medical condition that could be expected to progress, recur, or change to such an extend that it may bias the assessment of the clinical status of the patient to a significant degree or put the patient at special risk;
24. Ocular disorders in the study eye that may confound interpretation of study results, compromise visual acuity or require medical or surgical intervention during the 6 month study period, including cataract, retinal vascular occlusion, retinal detachment, macular hole, or choroidal neovascularisation of any cause (e.g., AMD, ocular histoplasmosis, or pathologic myopia);
25. Prior episode of RVO;
26. Evidence on examination of sight-threatening diabetic retinopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Estimated)
Dates: Start 2012-06; Primary Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Best corrected visual acuity | 6 months
  The primary outcome is the change in best-corrected visual acuitiy (BCVA) in the study eye from baseline to month 6 assessed with EDTRS-like VA charts at an initial distance of four meter.

SECONDARY OUTCOMES:
Proportion of patients with a gain or loss of 15 letters or more | 6 months
  The proportion of patients with a gain or loss of 15 letters or more at 6 months compared to baseline BCVA
Change in leakage on fluorescein angiography | 6 months
  The change in leakage on fluorescein angiography at the 6 month exit visit compared to baseline
Change in foveal thickness by optical coherence tomography | 6 months
  The change in foveal thickness (central area thickness) by optical coherence tomography at 6 months compared to baseline
The number of adverse events | 6 months
  The number of adverse events that occurred in the time frame of 6 months and a classification of the type of adverse events
Costs per quality adjusted life-year of the two treatments | 6 months
  The costs per quality adjusted life-year of the two treatments, results will be based on the use of standardized health questionnaires (EQ5D or HUI3)
The proportion of patients with a BCVA of 20/40 or more | 6 months
  The proportion of patients with a BCVA of 20/40 or more at 6 months compared to baseline BCVA

CONTACTS AND LOCATIONS:
Overall Officials: Reinier O Schlingemann, MD, PhD, Principal Investigator — Academic Medical Center, Dept. Ophthalmology, Room A2-122, Meibergdreef 9, 1105 AZ Amsterdam, The Netherlands
Locations (1):
- Academic Medical Center, Dept. Ophthalmology, Amsterdam, Netherlands